CLINICAL TRIAL: NCT02056314
Title: Developing and Evaluating Effectiveness of a Reinstatement Tutorial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Lottery and Gaming (Unknown)
Responsible Party: Principal Investigator, Nigel Turner, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 126/2013
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Problem Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- brochure (Active Comparator): The participants will be given a brochure that describes problem gambling and recommends methods of staying in control of gambling such as coping skills.
  Interventions: Other: brochure
- electronic tutorial (Experimental): The participants will be given an electronic tutorial that will explain how to stay in control of their gambling including information about coping skills, warning signs, and information about myths related to gambling.
  Interventions: Other: electronic tutorial

INTERVENTIONS:
Other: electronic tutorial — The electronic tutorial will provide information to the participants about the nature of gambling, and how to protect themselves against the risks of problem gambling including information on coping skills, and myths associated with gambling.
  Arms: electronic tutorial
Other: brochure — The brochure is the current means of informing people about the risks of problem gambling. It includes information about problem gambling and help resources.
  Arms: brochure

SUMMARY:
This study will compare a computerized tutorial to a brochure in terms of their education impact of people who wish to end voluntary self-exclusion. Voluntary self-exclusion is a program used by people who seek to bar themselves from further access to the casino or other gambling venue. The Centre for Addiction and Mental Health (CAMH), in cooperation with Ontario Lottery and Gaming (OLG), is developing a tutorial designed to provide practical information to players who choose to reinstate and return to gambling. The goal of this study is to determine if this new computerized tutorial decreases the harm of gambling experienced by gamblers who are reinstated. For example, are they less likely to relapsing to problematic levels of gambling.

DETAILED DESCRIPTION:
Voluntary self-exclusion is a program used by people who seek to bar themselves from further access to the casino or other gambling venue. Currently there are over 10000 people in the program. Although some self-exclusion programs place a permanent ban on the individual, others offer the possibility of reinstatement after a period of time. Many problem gamblers actually do change their minds about self-exclusion and wish to return to gambling. Centre for Addiction and Mental Health (CAMH), in cooperation with Ontario Lottery and Gaming (OLG), is developing a tutorial designed to provide practical information to players who choose to reinstate and return to gambling. The goal of this study is to evaluate an the intervention to determine its impact on problem gamblers who is reinstated from relapsing to problematic levels of gambling. The content for the tutorial will be informed by CAMH, will be developed for land based gambling, and also adapted for online gambling as well.

ELIGIBILITY:
Inclusion Criteria:

* people currently in the voluntary self-exclusion program who wish to be reinstated (allowed back into the casino to gamble).

Exclusion Criteria:

* people who are not currently in the voluntary self-exclusion program

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-02; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Gambling frequency | 6 months
  The frequency with which the person is gambling will be used to determine if they are gambling problematically.

SECONDARY OUTCOMES:
Gambling cravings | 6 months
  This will be measured using the Gambling Symptom Assessment Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel E. Turner, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada